CLINICAL TRIAL: NCT05649800
Title: Evaluating the Feasibility of Remote Haemodynamic Monitoring in a Cohort of Multi-ethnic Chronic Stroke Patients Using a Novel User Interface and Artificial Intelligence Algorithms
Brief Title: Vascular mEchanisms in, Stroke, dePression, dementiA, and deliRum: The VESPAR Project
Acronym: VESPAR
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0872
Record Dates: First submitted 2022-11-22; First posted 2022-12-14 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Dysfunction; Stroke; Dementia; Depression; Delirium
MeSH Terms: conditions — Cognitive Dysfunction; Stroke; Dementia; Depression; Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Healthy: Healthy adults ages over 65 years
- Stroke: Stroke patients aged over 65 years
- Dementia: Dementia patients aged over 65 years
- Depression: Depression patients aged over 65 years
- Delirium: Delirium patients aged over 65 years

SUMMARY:
The goal of this observational study is to determine the feasibility of using integrated Transcranial Doppler Ultrasonography or Near Infrared Spectroscopy to detect changes in cerebral autoregulation and neurovascular coupling in healthy, stroke, dementia, depression and delirium populations. We also aim to:

* Determine the optimal stimulus for neurovascular coupling
* To derive sample size estimates for a future study
* To develop a multilevel, multivariate model that can be applied to future datasets

DETAILED DESCRIPTION:
Healthy participants and those with dementia or depression will be invited to one assessment in the Cerebral Haemodynamics in Ageing and Stroke Medicine (CHiASM) research laboratory based at the Leicester Royal Infirmary. For participants with delirium, this assessment will be carried out on the ward to minimise changes to their environment. For participants with stroke, an assessment will be made by LB or JM as to whether it is most appropriate to undertake the study assessment in the lab or on the ward. Capacity will be assessed in compliance with the provisions of the Mental Capacity Act (England and Wales) 2005 to ensure full consent can be given by the potential research participant.

Participants will under-go two recordings of continuous beat-to-beat cerebral blood flow velocity (CBV) using transcranial Doppler ultrasonography (TCD), blood pressure (BP) using a Finometer, end-tidal CO2 (EtCO2) using nasal capnography, heart rate (HR) using a 3-lead ECG, and cortical oxygenation via pre-frontal near-infrared spectroscopy (NIRS). The first recording will last 5 minutes and will be conducted at rest. The second recording will last approximately 15 minutes and use four stimulation paradigms (cognitive, motor, sensory, and visual).

At the end of the cerebrovascular assessment, participants will be asked to complete questionnaires formally assessing cognitive function (Montreal Cognitive Examination - MoCA), mood (Geriatric Depression-Scale 15 - GDS-15), and delirium (4AT), where these weren't conducted as part of the screening process. Stroke patients will undergo additional scales to assess stroke severity (National Institute of Health Stroke Scale [NIHSS]) and dependency (modified Rankin Scale [mRS]).

Balance and community monitoring sub-study Suitable participants will be invited to undergo an additional or separate assessment on integrated TCD-NIRS during a balance assessment that assesses postural sway in different conditions. These include with visual input or standing on foam with and without the eyes open Participants in the balance sub-study will undergo additional measurements of lying and standing BP, and a fall assessment (Falls Efficacy Scale International [FES-I]). All participants will be offered an optional follow-up using Infiniwell remote monitoring systems (Lifesignals© Biosensor https://lifesignals.com/wearable-biosensors/1ax-biosensor/) in the community.

Follow-up assessment Participants with a diagnosis of stroke or delirium will be asked to return at 3 months for a follow-up neurovascular assessment (identical to the first). Only the stroke and delirium groups are being asked to return at follow-up as these two conditions are likely to improve over time.

ELIGIBILITY:
* Inclusion Criteria:
* Healthy adults aged over 65 years, free from medical comorbidities or medications that can adversely affect cognitive function or cerebral haemodynamics;
* Stable, well controlled comorbidities (e.g. hypertension);
* A diagnosis of dementia (major neurocognitive disorder), depression, or delirium, according to the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-V) criteria;
* Participants on or off anti-dementia drug therapy (acetylcholinesterase inhibitors, NMDA receptor antagonists), and antidepressants;
* A diagnosis of ischaemic (IS) or haemorrhagic (ICH) stroke according to clinical and/or radiological findings, within 72 hours of symptom onset
* Exclusion Criteria:
* Poorly controlled medical comorbidities affecting cerebral haemodynamics or cognitive function (e.g., heart failure, hypertension, type two diabetes);
* Clinically unstable or too unwell to cooperate with the study protocol;
* Lacks capacity or personal consultee to consent to the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Healthy and Stroke, Dementia, Depression and Delirium Individuals aged over 65 years
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-11-26 (Actual); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Good quality TCD-NIRS data | 3 years
  Number and percentage of complete TCD-NIRS assessments with good quality data (above the upper 95% confidence limit for the mean square error of the sample for at least one parameter) across all consented participants.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jatinder Minhas, Principal Investigator — Clinical Associate Professor of Stroke Medicine
Locations (2):
- United Kingdom (2):
  - University Hospitals of Leicester NHS Trust, Leicester, Leicestershire
  - Leicestershire Partnership Trust, Leicester, Leicestershire

IPD SHARING:
Plan to Share IPD: No